CLINICAL TRIAL: NCT07130656
Title: A Novel AI Algorithm With Enhanced Accuracy for Surveillance of Deep Surgical Site Infections After Elective Colorectal Surgery. A Diagnostic Accuracy Study.
Brief Title: AI Algorithm for Surveillance of Deep Surgical Site Infections After Elective Colorectal Surgery.
Acronym: Infect-IA-2
Status: Recruiting | Type: Observational
Sponsor: Hospital de Granollers (Other)
Responsible Party: Principal Investigator, Josep M Badia, Prof, Hospital de Granollers
Other Study IDs: Infect-IA-2
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Surgical Site Infection
Keywords: Surgical Site Infection; Surveillance; Articicial inteligence; Algorithms
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients assessed for SSI using the standard manual surveillance method: Patients undergoing colorectal surgery enrolled in the nationwide SSI surveillance programme and assessed for SSI using the standard manual surveillance method.
  Interventions: Diagnostic Test: Diagnosis of SSI
- Patients assessed for SSI by an algorithm: Patients undergoing colorectal surgery enrolled in the nationwide SSI surveillance programme and assessed for SSI using the new algorithm
  Interventions: Diagnostic Test: Diagnosis of SSI

INTERVENTIONS:
Diagnostic Test: Diagnosis of SSI — Diagnosis of SSI by manual system in colorectal surgery procedures enrolled in the SSI surveillance programme.

SUMMARY:
Epidemiological surveillance is one of the eight core components of the World Health Organization Infection Prevention and Control Programmes. These include surveillance programmes for surgical site infection (SSI).

At present, for SSI surveillance, infection control teams perform a manual time-consuming work, which could make a transition to automated surveillance leveraging the new information technology.

The aim of this study was to evaluate the performance of a novel algorithm to detect SSI in a cohort of elective colorectal surgery patients who have been previously screened within a nationwide healthcare-associated infection surveillance system.

DETAILED DESCRIPTION:
Healthcare-associated infections (HAIs) have a negative impact on patient health, represent a significant healthcare and economic burden on healthcare systems and are considered the most preventable cause of serious adverse events in hospitalised patients.

Epidemiological surveillance is one of the eight core components of the World Health Organization (WHO) Infection Prevention and Control Programmes. These include surveillance programmes for surgical site infection (SSI), which have proven to be effective in all types of surgery and in a variety of settings.

For a programme to be effective, surveillance for HCAIs must be active, prospective and continuous, comprising a surveillance period up to 30-90 days post-intervention, to cover the high rate of SSIs detected after discharge.

At present, infection control teams perform a manual, prospective, time-consuming and almost artisanal work, which should make a transition to automated or semi-automated surveillance that leverages the possibilities offered by today's information technology.

The evolution of surveillance systems should benefit from this new possibilities offered by artificial intelligence, allowing automated detection of suspected SSI adverse events from clinical course text, microbiology reports or coding of diagnoses, procedures, complications and readmissions.

The aim of this study was to evaluate the performance of a novel algorithm to detect to detect SSI at its three anatomical levels, in a cohort of elective colorectal surgery patients who have been previously screened within a nationwide healthcare-associated infection surveillance system.

ELIGIBILITY:
Inclusion Criteria:

* Elective colorectal resection

Exclusion Criteria:

* Emergency surgery
* Infection present at operation
* Previous intestinal stoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective colorectal surgery in Hospital General de Granollers in the period 2010-2023
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Rate of surgical site infection | 30 days
  Rate of Surgical site infection according to the definitions of the CDC-NHSN (Centers for Disease Control and Prevention-National Healthcare Safety Network)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Navarro, PhD, Study Chair — Hospital General de Granollers
Locations (1):
- Hospital General de Granollers, Granollers, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casanova-Portoles D, Badia JM, Forero CG, Sanchez-Martinez N, Romero M, Alonso-Solis T, Limon E, Pujol M, Sancho J. A structured-data algorithm for semiautomated surveillance of surgical site infection after colorectal surgery: A diagnostic accuracy study. J Infect Public Health. 2026 Jan 15;19(4):103151. doi: 10.1016/j.jiph.2026.103151. Online ahead of print. PMID 41637931